CLINICAL TRIAL: NCT02627612
Title: Evaluation of ProVetus/Sponsorship Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-225
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Posttraumatic Stress Disorder; Reintegration; Social Support
Keywords: veteran; mentorship; Iraq/Afghanistan; treatment; PTSD; Suicide; Criminal Activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide | interventions — RID

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TM RWB PLUS Pro Vetus (Experimental): Research participants will receive an introductory email from the research team informing them that they were randomly assigned to this group and request that they voluntarily join TM RWB and receive mentorship from their matched and assigned mentor. In addition to TM RWB membership, research participants will also receive approximately four months of mentorship from a ProVetus mentor to assist them in further transitioning within the five domains.
  Interventions: Behavioral: Pro Vetus; Behavioral: Team Red, White, and Blue (TM RWB)
- TM RWB ONLY (Active Comparator): Research participants will receive an introductory email from the research team informing them that they were randomly assigned to this arm and request that they voluntarily join TM RWB. Weekly emails will provide lists of voluntary physical/social activities available to all Chapter members. No participation is required in these activities.
  Interventions: Behavioral: Team Red, White, and Blue (TM RWB)
- Control Group (Waitlist) (No Intervention): Research participants (recent Veterans) will be placed on a waitlist for approximately sixteen months. Based on their desires, the research participants in this group will have opportunity to belong to TM RWB plus receive approximately four months of mentorship from trained, peer-mentors (who are TM RWB volunteers).

INTERVENTIONS:
Behavioral: Pro Vetus — Volunteer mentors (a mix of Veterans and non-Veterans) in the civilian community work with transitioning Veterans for approximately four months within five transition domains (1. Employment/Education, 2. Housing, 3. Family and Legal, 4. Social/Community/ Physical Fitness and 5. Medical Care).
  Arms: TM RWB PLUS Pro Vetus
Behavioral: Team Red, White, and Blue (TM RWB) — TM RWB is a 501(c)(3) non-profit, Veteran support organization found in 2010. Its mission is to enrich the lives of America's Veterans by connecting them to their community through physical and social activity. Central to TM RWB's mission is that inspiring Veterans to become physically active will create opportunities to establish authentic connections to other Veterans, active duty military, and civilians as well as improve the chances for continued successful integration. Enrollment in TM RWB takes place by simply signing up online and providing a name, email address, and zip code (teamrwb.org). TM RWB is not designed as a mental health intervention.
  Arms: TM RWB ONLY; TM RWB PLUS Pro Vetus

SUMMARY:
Some Veterans who recently served in the military report significant psychological problems based on their experiences in the military. Stressors that these Veterans face when they transition out of the military can acerbate these problems and negatively impact their long-term physical and psychological well-being. The investigators are conducting a randomized controlled trial to evaluate the efficacy of providing Veterans who are transitioning back into their civilian communities trained, peer mentorship (Pro Vetus) and membership in a Veteran Support Organization (VSO) Team Red, White, and Blue (TM RWB) to reduce transition stressors, maintain psychological and physical health, reduce suicides and reduce criminal incidents.

DETAILED DESCRIPTION:
The evidence basis suggests that the pre-existing psychological states of those who enter the military, compounded by combat exposure, may further deteriorate with the loss of leadership and social support by leaving the structured military environment. In a perfect situation, practitioners could simply track these "at risk" individuals throughout their military service and then ensure that they received medical services through the Veterans Affairs after transitioning to the civilian sector. It would appear that such an approach would help to reduce suicide in Veterans since studies have shown that Vietnam Veterans with a posttraumatic stress disorder (PTSD) diagnosis approximately forty years after Vietnam (i.e., worsening chronic or high-stable) were almost 3 times more likely to have a suicide attempt compared to Veterans without PTSD. Additionally, the suicide rate for Veterans who actually do seek VA healthcare services has improved in recent years (approximately 34 per 100,000 in 2008 to approximately 28 per 100,000 in 2010). This is a testament to the services that the VA is providing Veterans who seek care.

Unfortunately, this approach has not been fully successful for two reasons. First, many of the transitioning Veterans who need services the most will not seek these services primarily because of the prevalent stigma against mental health services among Veterans. For example, previous research found that only 34 percent of National Guard Veterans who screened positive for PTSD after a deployment to Afghanistan actually sought treatment within their first year after redeploying home and transitioning back into the civilian sector. It is important to note that of the 1.7 million Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans eligible for Veteran Affairs (VA) services that only 58 percent (998,004) have ever utilized these services. Second, such an approach does not take into consideration the cumulative impact upon Veterans of losing the protective factors of leadership and social support after they transition into the civilian sector and the compounding effect of transitioning stressors upon Service Members. For example, it is possible that some Veterans could be within a low-stable or resilience trajectory while experiencing the protective factors of leadership and social support in the military but then worsen after these factors dissipate and transitioning stressors take effect. In fact, a longitudinal study of National Guard Service Members ascertained the impact of transitioning stressors (i.e., issues with employment or financial difficulties, issues related to housing, and issues related to marital and family problems) upon Veterans returning from combat and transitioning back into the civilian sector. The study found that transitioning stressors were highly correlated with psychological problems (i.e., PTSD, depression and alcohol dependence) and were more associated with suicidal ideation than each of the psychological problems. In fact, after adjusting for individual psychological problems, the odds of suicidal ideation among Veterans experiencing the highest number of transitioning stressors were 5.4 times that of Veterans experiencing no transitioning stressors. Additionally, Service Members who experienced a divorce after deployment were at an even greater risk for suicidal ideation. The impact of transitioning stressors may help to explain why 96 percent of a sample of 754 OEF/OIF Veterans who sought care from the VA (between 2003 and 2007) expressed interest in receiving services or information concerning transitioning problems. The most frequently reported interests were related to Veteran Affairs benefits (83 percent of those surveyed) and schooling, employment, or job training (80 percent of those surveyed).

These two reasons together may help to explain why the suicide rate for Veterans who do not seek services from the VA, after transitioning into the civilian sector, has risen within the last few years from approximately 34 per 100,000 in 2008 to approximately 39 per 100,000 in 2010. It appears that those most at risk are our youngest Veterans (18-24 year olds). The suicide rate for young Veterans who used VA services spiked from 46.1 per 100,000 in 2009 to 79.1 per 100,000 in 2011. The investigators assume that the rate for our young Veterans who haven't ever used VA services is even significantly higher. This means that among the 42 percent (726,054) of OEF/OIF Veterans who haven't ever used services could possibly be the riskiest Veterans for suicide. This is a major concern of ours and constitutes what this research study refers to as the "Deadly Gap", which consists of the time between military service for a Veteran and their successful transition back into the civilian sector.

In trying to develop an intervention that addresses the concerns listed above, the investigators reviewed already established programs within the military and successful programs within the civilian sector. Of note, the investigators referenced the "Best Practices Identified for Peer Support Programs" published by the Defense Centers of Excellence for Psychological Health & Traumatic Brain Injury (TBI). Additionally, the U.S. Army provides a mentor/sponsorship program (i.e., Total Army Transition Program) that assists every Soldier to successfully navigate a Permanent Change of Station during which time a Soldier transfers from one Army base to another. In this existing program, the sponsor ensures that the Soldier transfers to the next duty station within such critical domains as--employment/duty, housing, family, social/community/ physical activities, and medical care. The sponsor doesn't provide services within each of these domains but instead guides the transferring Soldiers and connects him or her to the organizations/individuals which do provide these services. Unfortunately, no comprehensive system currently exists to enable Service Members to execute their transition from the military to the civilian sector (or "Expiration Term of Service"). The stressors that can result from transitions within any of the domains can accumulate and acerbate pre-existing physical or psychological concerns, especially suicide. The lack of such a program forces some transitioning Service Members to navigate the "deadly gap" by themselves.

The investigators were also drawn to the successes of some programs for OEF/OIF Veterans at institutions of higher learning. For the institutions that have been successful in transitioning Veterans into academic life, it appears that they have focused on continuing informal and formal leadership for the Veterans by--emphasizing positive interactions with faculty and support personnel, providing peer mentors, establishing a social support structure for the Veterans through connecting new Veteran students with other Veterans on campus, and creating a cooperative network of Veteran service agencies (especially with the VA) aimed at easing the transition for Veterans. It appears that such deliberate and synchronized interventions are effective because they maintain positive protective factors-leadership and social support-for transitioning Service Members and help to minimize transitioning stressors. The investigators saw the opportunity to leverage the existing informal social network established by the New York City Chapter of TM RWB to test a new intervention, Pro Vetus. It capitalizes on the existing informal social support network created by TM RWB, with the added intervention of formal social support and resources through trained leadership provided by Pro Vetus.

With all of the above information, the investigators designed Pro Vetus upon the following five principles to bridge the deadly gap:

1. Focused on Successful Transition of OEF/OIF Veterans to enable them to become the next corporate and societal leaders (It is not an intervention based on a medical model of treating disorders).
2. Focused on maximizing protective factors of leadership and social support for all transitioning Veterans. Everyone could benefit from a trained mentor to assist in navigating the "deadly gap."
3. Focused on short-term transition of Veterans to the civilian sector within the five domains (employment/education, housing, family, social/community/physical activity, and medical care)
4. Focused on establishing a supportive and collaborative environment for all agencies that serve Veterans facilitated by capabilities provided by Unite Us and Google.
5. Focused on mentors establishing positive interpersonal relationships with recently transitioned Veterans and their family members; Mentors are trained to provide "Buddy Aid" (if necessary) and immediately connect Veterans to necessary services. Mentors receive support from team leaders and the Department of VA Suicide Prevention Coordinators to ensure they provide the best support possible to transitioned Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over, prior military service within the last twelve years, and currently reside within the NYC area (and anticipate staying within the area for at least one year) or will move to NYC area prior to December 2016 (and anticipate staying for at least one year).

Exclusion Criteria:

* Previous membership within Team Red, White, and Blue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in baseline PCL (PTSD) scores across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Military to Civilian Questionnaire scores across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Social Support Scale scores across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline suicidality across 2 timepoints | 16 months after baseline and 5 years after baseline
  Outcome measured through Mortality (Suicide) Data Center for Disease Control

SECONDARY OUTCOMES:
Change in baseline Veteran Rand 36 scores across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline PHQ-15 scores across 3 time points | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Criminal Background Record across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Criminal Background Self-Report across 3 timepoints | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline AUDIT-C (Alcohol Use) scores across 3 time points | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Quality of Life, Enjoyment and Satisfaction scores across 3 time points | Baseline, 3 months after, 10 months after, 16 months after
Change in baseline Social Adjustment Scale scores across 3 time points | Baseline, 3 months after, 10 months after, 16 months after

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Geraci, LMHC, Principal Investigator — Teachers College, Columbia University; George Bonanno, PhD, Study Chair — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No